CLINICAL TRIAL: NCT04333849
Title: Telephony Or Videophony for Isolated elDerly in Maine-Et-Loire 49 During COVID-19
Acronym: TOVID-49
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2020/29
Record Dates: First submitted 2020-04-01; First posted 2020-04-03 (Actual); Last update posted 2020-07-20 (Actual); Status verified 2020-03

CONDITIONS: Coronavirus
MeSH Terms: conditions — Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current health crisis at COVID-19 is forcing us to profoundly rethink our social organizations, especially towards our most fragile seniors. Prohibitions on visits to Nursing Homes and care services, although essential to control the epidemic, are also becoming a major source of social isolation and loneliness for these fragile populations. The only source of residual social ties during a period of confinement remains dematerialised communication via the various existing communication channels (in particular telephone calls or video telephony).

As soon as the COVID-19 crisis began and the first visiting restrictions were imposed on patients in the geriatric department of the Angers Univesity Hospital and the Retirement Home / long-term care unit, acute care geriatric unit of Angers offered patients and residents the opportunity to organize communication with their relatives via videophone calls. Initial feedback from the field shows us that, contrary to our intuition, patients and residents are not necessarily asking for communication to the outside world and, when they are, the preferred channel is not necessarily video telephony but often a simple phone call with relatives. Even though the vast majority of projects aimed at setting up communication aids for the elderly now rely on videophonic support, these initial observations in everyday care situations raise questions about the directions taken in this area. Also, the investigators ask themselves the following question: in the absence of a physical meeting, what is the preferred means of communication for elderly people in isolation in hospital or in Retirement Home? This study will make it possible to propose the most appropriate solutions for breaking isolation for the hospitalized or institutionalized geriatric population in order to limit as much as possible the increase in social isolation imposed by restrictions on movement during epidemics.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalisation in the acute care geriatric unit (Angers UH) or institutionalization in St Nicolas during the isolation measures linked to the SARS-CoV-2 epidemic.

Exclusion Criteria:

* Refusal to participate.
* Contraindication posed by the medical team to proposing dematerialized communication.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients are recruited during their hospitalisation in acute care geriatric unit or institutionalization in St Nicolas during the isolation measures linked to the SARS-CoV-2 epidemic.
Sampling Method: Probability Sample
Enrollment: 132 (Actual)
Dates: Start 2020-03-25 (Actual); Primary Completion 2020-05-11 (Actual); Study Completion 2020-05-11 (Actual)

PRIMARY OUTCOMES:
Preferred means of communication for elderly people in isolation, hospitalized in the acute care geriatric unit or residing at St Nicolas nursing home (Angers UH). | at baseline (day 0)
  Choice between videophony, telephony or neither.

SECONDARY OUTCOMES:
proportion of elderly people with loss of functional independence to communicate with their relatives. | at baseline (day 0)
  Aid received or not (by a caregiver) in connecting with the relative.
level of satisfaction of patients who have benefited from a telephone call. | at baseline (day 0)
  The satisfaction will be assessed using a non-validated satisfaction questionnaire based on a forced choice Likert scale in 6 points from 1 to 6. Patients will be considered as satisfied if the mean score is over 4 on 6.
level of satisfaction of patients who have benefited from a videophone call. | at baseline (day 0)
  The satisfaction will be assessed using a non-validated satisfaction questionnaire based on a forced choice Likert scale in 6 points from 1 to 6. Patients will be considered as satisfied if the mean score is over 4 on 6.
satisfaction level of older people according to the means of communication used. | at baseline (day 0)
  The satisfaction averages of the two groups wishing to use a means of communication (telephony or videophony) will be compared by a Student t-test.
impact of age on the preferred means of communication. | at baseline (day 0)

CONTACTS AND LOCATIONS:
Locations (1):
- Angers University Hospital, Angers, France

REFERENCES:
- [Derived] Sacco G, Lleonart S, Simon R, Noublanche F, Annweiler C; TOVID Study Group. Communication Technology Preferences of Hospitalized and Institutionalized Frail Older Adults During COVID-19 Confinement: Cross-Sectional Survey Study. JMIR Mhealth Uhealth. 2020 Sep 18;8(9):e21845. doi: 10.2196/21845. PMID 32896832